CLINICAL TRIAL: NCT06726707
Title: COPPER: An Adaptative Design, Randomized, Multicenter, Controlled, Double-Blinded Exploratory Trial, Evaluating the Management of Incontinence-Associated Dermatitis Using Copper Containing Absorbing Incontinence Products
Brief Title: COPPER: A Trial Evaluating Copper-based Products for Incontinence-associated Dermatitis
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: At the discretion of the sponsor
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Essity Hygiene and Health AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COPPER_Trial
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Incontinence-associated Dermatitis
Keywords: urinary incontinence; fecal incontinence; copper
MeSH Terms: conditions — Urinary Incontinence; Fecal Incontinence

STUDY DESIGN:
Intervention Model Description: Adaptative Design, Randomized, Multicenter, Controlled, Double-Blinded Exploratory trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Copper-based product (Experimental): Individuals enrolled in the treatment with diapers embedded with a copper-based product plus usual care
  Interventions: Combination Product: Diaper with a copper-based product + usual care
- Control (Active Comparator): Individuals enrolled in the treatment with common diapers plus usual care
  Interventions: Combination Product: Barrier product with common diaper

INTERVENTIONS:
Combination Product: Diaper with a copper-based product + usual care — The intervention is an incontinence aid product and its performance is related to its ability to absorb and contain urine/ feces as well as keeping the skin dry.
  Arms: Copper-based product
Combination Product: Barrier product with common diaper — The common diaper is an incontinence aid and its performance is related to its ability to absorb and contain urine/ feces as well as keeping the skin dry.
  Arms: Control

SUMMARY:
As there are currently no evidence on the benefit of absorbing incontinence products with copper to stabilize IAD in the elderly, thus, this study will assess the capacity and safety of an absorbing incontinence products with a copper-based substance for the management of adults with incontinence-associated dermatitis, compared to an absorbing incontinence products with no substance. This approach may contribute for IAD management arsenal, since clinical evidence on the efficiency of products available in the market to manage IAD is frail, as seen in systematic reviews mentioned above. We believe copper, as a barrier product, has the potential to perform well in this clinical setting of IAD, as it performed well in other settings.

DETAILED DESCRIPTION:
This study adopts an exploratory trial design with an adaptive approach. It is randomized, multicenter, controlled, and double-blinded, with parallel groups and blinded outcome adjudication. The study hypothesis suggests that incontinence products infused with copper-based substances may provide superior stabilization of IAD compared to control products.

The primary objective of the study is to evaluate the effectiveness of absorbing incontinence products containing a copper-based substance in stabilizing incontinence-associated dermatitis (IAD) in adults with moderate to severe urinary and/or fecal incontinence. This will be compared against standard absorbing incontinence products without copper-based substances, with both groups receiving usual care. Secondary objectives include assessing improvements in pain within 14 and 28 days, evaluating quality of life improvements over 28 days, and measuring changes in skin health scores from baseline to 14 and 28 days.

Participants will be adults aged 60 years or older, experiencing moderate to severe urinary and/or fecal incontinence. Eligibility will be determined using specific scales outlined in the study rationale. Recruitment will target individuals in long-term care facilities or hospital wards located within São Paulo municipality and its metropolitan area in Brazil. Feasibility assessments will be conducted at each site during an initial visit. Sites deemed suitable will then proceed with participant recruitment.

This study seeks to address critical aspects of managing IAD, particularly through innovative copper-based products. By focusing on clinical endpoints such as pain reduction, quality of life enhancements, and improvements in skin health, the trial aims to provide evidence supporting the potential benefits of copper-infused incontinence products over traditional alternatives.

ELIGIBILITY:
Inclusion Criteria:

* Ability and capability to participate in the study and follow study procedures as determined by the investigator.
* With moderate or more intense urinary (ISI ≥ 3) and/or fecal incontinence (Pescatori et al. (B1, B2, B3, C1, C2, C3);
* Current users of absorbing incontinence products.
* Diagnosed with incontinence-associated dermatitis GLOBIAD 1A or 2A.

Exclusion Criteria:

* Incontinence-associated dermatitis GLOBIAD 1B or 2B;
* The subject who knows about allergy or a history of an adverse reaction to product ingredients or to any topical preparations or skincare products;
* The subject who has an active skin condition or a history of recurrent skin conditions, except IAD, that may affect IAD healing;
* The subject who was treated in the previous week with systemic or topical agents (except for IAD) that may affect IAD healing process (e.g., steroids);
* Subject with a score < 10 in Mini Nutritional Assessment - Short Form;
* Subjects with diabetes.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of non-progressing IAD 14 days | 14 days
  Proportion of non-progressing IAD after 14 days from randomization start by GLOBIAD criterion.

SECONDARY OUTCOMES:
Proportion of non-progressing IAD 28 days | 28 days
  Proportion of non-progressing IAD after 28 days from randomization start by GLOBIAD criterion.
Pain assessment | 14 and 28 days
  Pain assessment using the numerical scale in 14 and 28 days; the scales goes from 0, for no pain, to 10, for the worst pain ever felt by the patient.
Quality of life SF12 | 28 days
  Quality of life assessment in the 28th day (Short-Form 12 Health Survey). The maximum score is 100, and the higher the better.
Skin health by skin health assessment tool | 14 and 28 days
  The skin health of the subjects after 14 and 28 days using the skin health assessment tool, a visual assessment tool with no ordinal scale.
Time to resolution of IAD | From enrollment to resolution, mean of 4 to 7 days
  Time to resolution of IAD
Reoccurrence of IAD | From resolution of the first episode of IAD to the 28th day
  Reoccurrence of IAD during the follow-up of 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Henrique A Rodrigues da Fonseca, PhD, Principal Investigator — Hospital Israelita Albert Einstein - ARO

IPD SHARING:
Plan to Share IPD: No